CLINICAL TRIAL: NCT05373342
Title: Feasibility Study to Evaluate the Role of a Novel Device in the Prevention of Retained Items In Childbirth Environment- Clinical Usability Pilot Study
Brief Title: Feasibility Study to Evaluate the Role of a Novel Device in Childbirth
Acronym: PRINCE
Status: Not yet recruiting | Type: Observational
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021SUR119
Record Dates: First submitted 2022-05-03; First posted 2022-05-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Surgical Item, Retained; Childbirth
MeSH Terms: conditions — Foreign Bodies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- iCount Device: A novel external device which can count the swabs and surgical tampons used during childbirth in an objective and validated manner.
  Interventions: Device: iCount system assembled with swabs
- User Feedback Survey: Feedback will be taken from 20 users including midwives/ doctors.
  Users will be emailed an online survey or given the same survey as a printout to complete.
  All 20 users will also then also be approached to have a semi-structured interview.
  10 of the users who first express interest will be interviewed.

INTERVENTIONS:
Device: iCount system assembled with swabs — Designed as single use. Intended purpose - To be used to count swabs and tampons after childbirth in an objective manner. This is intended to be used in women during and after childbirth.
  Groups: iCount Device

SUMMARY:
Accidentally retained surgical items or swabs are well-recognised errors that result in adverse consequences for patients. This error is one of the commonest "Never Events" - patient safety incidents that are considered preventable. Although uncommon, these incidents can have devastating consequences. Retained surgical items have 70% re-interventions, reaching 80% morbidity and 35% mortality.

Swabs or sponges are like small towels that soak up blood and body fluids so that the surgeon can visualise the operating area effectively. Swabs are used in all areas of surgery which include operations on the tummy, chest, limbs. They are also used in the vagina during childbirth, to assess for tears and to minimise blood oozing from the vagina.

The common risk factors for this error are out of hours surgical or childbirth procedures, multiple handovers in the care of the patient, raised BMI (Body Mass Index) and unplanned change to the operative intervention.

As the name suggests, a 'never event' should never happen in the first place. Never. Unfortunately, this is not the case. Incidents involving surgical swabs being left behind, particularly during a caesarean section or a perineal repair following a vaginal birth, are still happening despite over 100 years of institutional awareness of the problem and tentative solutions being implemented in clinical practice.

never-event incidents involving retained surgical swabs are a widespread problem affecting healthcare systems worldwide. It is therefore reasonable to ask the question: why are surgical swabs being left behind and what can be done to prevent this from happening?

ELIGIBILITY:
Inclusion Criteria:

* Midwifery lead and consultant lead patient older than 18 years.
* Consented to participation after an informed choice.

Exclusion Criteria:

• Under 18 years of age

Antenatal (before labour):

* Patients who have a high risk of expected/unexpected maternal, fetal or neonatal deterioration such that during birth, the focus of attention would be towards safe patient care and observation required for using the swab-counter device system would not be possible such as :
* Patients who are seriously unwell and require high dependency care.
* Maternal cardiac conditions
* Severe pre-eclampsia
* Fetal anomalies where neonatal deterioration is expected (These will be relatively rare conditions where the doctor/midwife would decide to not recruit the patient)

Intrapartum and postpartum factors:

* Patient having an emergency Caesarean section instead of a vaginal birth due to maternal or fetal indication.
* Eclampsia (seizure/fitting in labour or after delivery)
* Maternal cardiac conditions requiring high dependency care
* Severe sepsis requiring high dependency care
* Fetal anomalies where neonatal deterioration is expected

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women during labour
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Rate of device count accuracy (conspicuity of spotting a missing swab) measured via staff questionnaire feedback | 12 months
User experience about general look and feel and user satisfaction (overall perception) measured via staff questionnaire feedback | 12 months
User perception about the confidence about the accuracy of the count with use of the device and thoughts about intention to use, if available (functionality) measured via staff questionnaire feedback | 12 months
User perception about the ease of learning of how to use the device measured via staff questionnaire feedback | 12 months
User perception of how device works within current system measured via staff questionnaire feedback | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Aditi Desai, Principal Investigator — The Royal Wolverhampton NHS Trust